CLINICAL TRIAL: NCT05355740
Title: The Effect of Post-surgical Chlorhexidine Mouth Washing on the Sub-gingival Periodontal Microbiome; a Pilot Study
Brief Title: The Effect of Post-surgical Chlorhexidine Mouth Washing on the Sub-gingival Periodontal Microbiome A Pilot Study
Acronym: SUPEM1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Jacob Horwitz MD, Director-Graduate Program in Periodontology, Rambam Health Care Campus
Other Study IDs: 0694-21-RMB CTIL
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Periodontitis; Subgingival Plaque
Keywords: chlorhexidine; subgingival plaque
MeSH Terms: conditions — Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Corsodyl — Corsodyl (a chlorhexidine mouthwash) will be used to rinse the mouth for one minute with 10 ml twice daily during ten days after oral surgery
  Other Names: Chlorhexidine mouthwash

SUMMARY:
Prospective applicants who conform with inclusion and exclusion criteria will be accepted into the study and sign a consent form.

Visit 1: After initial screening a case report form (CRF) will be filled, including information regarding general health, medication, demographic, oral and dental information. Participants will be clinically examined and the following data will be collected prior to surgery: microbial collection, Plaque score (PS) , probing pocket depth (PPD), bleeding on probing (BOP) at selected non-surgical and surgical teeth. Surgery will be performed followed by discharge with a bottle of chlorhexidine mouthwash and written instructions on its usage. Visit 2: Ten days after surgery sutures will be removed and collected for microbial examination. Microbial collection will be performed at non-surgical and surgical sites. Adverse events will be recorded and participants will be discharged from the study.

DETAILED DESCRIPTION:
Microbial identification: periodontal samples will be collected by the GeneFiX™ Saliva DNA Microbiome Collection Device (Isohelix). DNA Extraction - the MagMAX Microbiome Ultra Nucleic Acid Isolation Kits (Termo Fisher). DNA yields and purity - measuring absorbance at 260 nm, A260/A280 and A260/A230 ratios with the Nano-drop 2000 spectrophotometer (Nanodrop products, Wilmigton,USA). Microbiome sequencing - target V4 region of 16s rRNA gene will be sequenced on the Ion Torrent S5 instrument (Thermofisher) and analysis will be performed with the ERGO 2.0 platform ( iGenbio). The investigators will perform comparisons of alpha and beta diversity before and after intervention, as well as differential abundance of the taxa.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Scheduled for periodontal/dental surgery without pre- and/or post-surgical antibiotic therapy

Exclusion Criteria:

* Pre-existing conditions that may affect the microbiome, including diagnoses of diabetes, malignancy, alcoholism, previous head and neck radiation therapy
* Pregnancy and breast-feeding
* Chronic medications that are known to affect periodontal tissues such as Ca channel blockers and phenytoin
* Antibiotic therapy within the previous 6 weeks
* Mouthwash therapy within the previous 2 weeks
* Known allergy to CM or any of its constituents
* Smoking >10 cigarettes/day

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for periodontal surgery/dental extractions at the Rambam Department of Periodontology
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
alpha and beta diversity | 10-14 days
  sub-gingival microbiome changes between pre- and post- mouthwash usage in non-surgical sites and in surgical sites

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Horwitz, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No